CLINICAL TRIAL: NCT06263959
Title: A Randomized, Double-blind, Placebo-controlled Phase IIa Clinical Study to Evaluate the Safety and Efficacy of GST-HG131 Tablets in Patients With Chronic Hepatitis B
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Akeylink Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GST-HG131-II-01
Record Dates: First submitted 2024-01-07; First posted 2024-02-16 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — GST-HG131

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Patiants on stable nucleos(t)ide analog (NA) therapy will be randomized 4:1 to receive repeat dose of either GST-HG131 (Dose 1) or placebo for 28 days.
  Interventions: Drug: GST-HG131; Drug: Placebo to match GST-HG131
- Cohort 2 (Experimental): Patiants on stable nucleos(t)ide analog (NA) therapy will be randomized 4:1 to receive repeat dose of either GST-HG131 (Dose 2) or placebo for 28 days.
  Interventions: Drug: GST-HG131; Drug: Placebo to match GST-HG131
- Cohort 3 (Experimental): Patiants on stable nucleos(t)ide analog (NA) therapy will be randomized 4:1 to receive repeat dose of either GST-HG131 (Dose 1 or 2) or placebo for 12 weeks.
  Interventions: Drug: GST-HG131; Drug: Placebo to match GST-HG131

INTERVENTIONS:
Drug: GST-HG131 — GST-HG131 will be administered.
Drug: Placebo to match GST-HG131 — Placebo to match GST-HG131 will be administered.

SUMMARY:
A randomized, double-blind, placebo-controlled Phase IIa clinical study to evaluate the safety and efficacy of GST-HG131 tablets in patients with chronic hepatitis B

ELIGIBILITY:
Inclusion Criteria:

1. Able to sign the informed consent form，and fully understand the test content, process and possible adverse reactions；
2. Males and females aged 35-65 ,able to complete research in accordance with test plan requirements;
3. Participants who have no childbearing plan in next year,and must agree to voluntarily use the contraceptive methods specified in the protocol from screening to 6 months after the last dose of the study；
4. The weight of male patients shall not be less than 50 kg, and the weight of female patients is not less than 45 kg. Body mass index (BMI = weight (kg)/height 2 (m2)) in the range of 18.0~35.0 kg/m2；
5. Participants who have received stable NA therapy for more than half a year and have maintained the NA regimen for ≥3 months prior to screening；
6. At least two tests within 28 days of the screening period (more than 1 week apart) with HBV DNA lower than LLOQ；
7. HBeAg negative, 100≤HBsAg quantitative ≤1500 IU/mL, serum ALT<1×ULN during screening;
8. The normal or abnormal results of vital signs assessment, physical examination and 12-lead electrocardiogram during the screening period and baseline period have no clinical significance；
9. Able to communicate well with clinical staff and complete the trial according to protocol requirements。

Exclusion Criteria:

1. Participants with a history of allergy to the any ingredient or excipients of the drug under study；
2. Patients who cannot tolerate venous blood collection and have a history of needle fainting or blood fainting；
3. Patients with major trauma or major surgery within 3 months before screening; or plan to have surgery during the study；
4. Blood donation or blood loss ≥400 mL within 3 months prior to screening, or received blood transfusion; or blood donation or blood loss ≥200 mL within 1 month prior to screening；
5. A history of alcohol or drug abuse or dependence；
6. Participants have participated in clinical trials of drugs or medical devices (except in vitro diagnostic reagents) within 3 months prior to administration；
7. Use of any hepatitis B drug other than NUC within 1 year prior to administration；
8. Participants with systemic use of immunosuppressants, immunomodulators (excluding interferon) and cytotoxic drugs within 6 months before screening; Or those who received live attenuated vaccine within 1 month before screening；
9. Participants with clinically significant acute or chronic liver disease caused by non-HBV infection who were judged by the investigator to be unsuitable for the study；
10. Participants with a history of cirrhosis (e.g., the subject had a histopathological examination of the liver and reported cirrhosis, or had an endoscopic examination indicating varicose esophagus and fundus veins);
11. Participants with hepatitis B cirrhosis in the confirmed or suspected decompensated stage, including but not limited to: hepatic encephalopathy, hepatorenal syndrome, esophageal and fundus variceal bleeding, spleen enlargement, ascites, primary liver cancer, etc；
12. Participants with malignancy or history of other malignancies within 5 years prior to screening (except cured basal cell or squamous cell carcinoma of the skin and carcinoma in situ of the cervix)；
13. The investigators determined the presence of impaired gastrointestinal function or gastrointestinal disease that might affect oral drug absorption, such as severe gastrointestinal disease (peptic ulcer, erosive or atrophic gastritis), partial gastrectomy, and gastrointestinal symptoms > grade 2 at the time of screening (e.g., nausea, vomiting, or diarrhea)；
14. Participants with suspected or confirmed acute infections within 2 weeks prior to randomization；
15. Laboratory examination: platelet count < 90 x 10^9 / L; White blood cell count <3.0 x 10^9 / L; Neutrophils absolute value< 1.3 x 10^9 / L; Serum total bilirubin >2 x ULN. Albumin< 30 g/L; Creatinine clearance ≤ 60 mL/min or less; Prothrombin time international standardization ratio (INR) >1.5；
16. Serum AFP (AFP) is greater than 50 ㎍ / L (or 50 ng/mL) or imaging suggest possible malignant liver placeholder；
17. Hepatitis C antibody positive, treponema pallidum antibody positive and rapid plasma reagin test (RPR) positive,AIDS antigen/antibody positive；
18. Breastfeeding women or those who have a positive pregnancy test at screening or baseline；
19. The investigator believes that there are other subjects who are not suitable for participating in this trial.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-12-26 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in HBsAg levels | Baseline and up to 56 days(Cohort1 and 2) or 16 weeks(Cohort3)
  Change from Baseline in HBsAg levels

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs), serious adverse events (SAEs), and withdrawals due to AEs | Up to 56 days(Cohort1 and 2) or 16 weeks(Cohort3)
  Number of participants with adverse events (AEs), serious adverse events (SAEs), and withdrawals due to AEs

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Medical Center of Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided